CLINICAL TRIAL: NCT05337553
Title: A Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of Taldefgrobep Alfa in Ambulatory and Non-Ambulatory Participants With Spinal Muscular Atrophy With Open-Label Extension
Brief Title: A Study to Evaluate the Efficacy and Safety of Taldefgrobep Alfa in Participants With Spinal Muscular Atrophy
Acronym: RESILIENT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV2000-301
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy; Neuromuscular Diseases; SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- taldefgrobep alfa (Experimental): taldefgrobep alfa - Double-blind (DB) Phase: Participants receive weight based 35 mg/50 mg weekly subcutaneous injection for 48-week DB phase.
  taldefgrobep alfa/taldefgrobep alfa - Extension Phase: Participants receive weight based 35 mg/50 mg weekly subcutaneous injection for Open label Extension (OLE) phase.
  Interventions: Drug: taldefgrobep alfa
- Placebo (Placebo Comparator): Placebo - Double-blind (DB) Phase: Participants receive weight based 35 mg/50 mg weekly subcutaneous injection for 48-week DB phase.
  Placebo/taldefgrobep alfa - Extension Phase: Participants who receive placebo during DB phase, receive weight based 35 mg/50 mg weekly subcutaneous taldefgrobep alfa injection for OLE phase.
  Interventions: Drug: Placebo; Drug: taldefgrobep alfa

INTERVENTIONS:
Drug: taldefgrobep alfa — DB Phase: 35 mg/50 mg weekly subcutaneous injection
  Other Names: BHV-2000; BMS-986089
  Arms: taldefgrobep alfa
Drug: Placebo — DB Phase: matching placebo 35 mg/50 mg weekly subcutaneous injection
  Arms: Placebo
Drug: taldefgrobep alfa — Extension Phase: 35 mg/50 mg weekly subcutaneous injection
  Other Names: BHV-2000; BMS-986089

SUMMARY:
This trial will study the efficacy and safety of taldefgrobep alfa as an adjunctive therapy for participants who are already taking a stable dose of nusinersen and/or risdiplam and/or have a history of onasemnogene abeparvovec, compared to placebo.

DETAILED DESCRIPTION:
Myostatin is a negative regulator of muscle growth. Blocking myostatin activity has been shown to increase muscle size and function. Taldefgrobep alfa directly blocks myostatin activity and was well tolerated in other clinical studies. In combination with medications that increase the amount of SMN protein in the body, taldefgrobep alfa has the potential to further improve motor function and clinical measures for people living with SMA.

ELIGIBILITY:
Key Inclusion Criteria:

* Spinal Muscular Atrophy confirmed by genetic diagnosis of 5q-autosomal recessive SMA as well as SMN2 copy number
* Ambulant or Non-Ambulant
* Treated with an SMA disease-modifying therapy and anticipated to remain on that same treatment regimen and dose throughout the trial including nusinersen and/or risdiplam and/or a history of onasemnogene abeparvovec

Key Exclusion Criteria:

* Cannot have previously taken anti-myostatin therapies
* Must weigh at least 15kg
* Respiratory insufficiency, defined by the medical necessity for invasive or non-invasive ventilation for daytime treatment while awake (use overnight or during daytime naps is acceptable)
* History of Spinal Fusion within 6 months of Screening. MAGEC rod nonsurgical adjustments are allowed during the study
* Presence of an implanted shunt for the drainage of CSF or an implanted central nervous system (CNS) catheter

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 269 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of taldefgrobep alfa compared to placebo in change in the 32 item Motor Function Measure (MFM-32) total score | Baseline to Week 48
  Change in MFM-32 total score from baseline to Week 48. Scores range from 0-3 on each item. The scores from the 32 items are summed and transformed to a 0-100 scale, with higher scores reflecting higher levels of functional abilities.

SECONDARY OUTCOMES:
Efficacy of taldefgrobep alfa compared to placebo in change in the Revised Upper Limb Module (RULM) score | Baseline to Week 48
  The RULM includes 20 items, graded from 0 to 2, with a maximum score of 37. Higher scores indicate better function.
Efficacy of taldefgrobep alfa compared to placebo in change in the Revised Hammersmith Scale (RHS) | Baseline to Week 48
  The RHS has a maximum score of 69 points (33 items are scored 0-2, and 3 items scored 0-1). Higher scores indicate better function.
Change from Baseline in lean body mass | Baseline, Week 48
  Body mass will be measured as change in kg (greater change meaning more improvement)
Change from Baseline in bone mineral density | Baseline, Week 48
  Bone mineral density will be measured by Z-score change (higher score indicates improvement)
Change from baseline in Tanner staging | Baseline, Week 48
Injection acceptability assessments | Week 48
  If local injection site reactions (such as redness, itching, swelling, hardening or bruising) are experienced, the acceptability is scored on a scale of 1-5 with 1 being totally acceptable and 5 being not at all acceptable If pain is experienced at the injection site, pain will be scored on a scale of 1-5 with 1 being totally acceptable and 5 being not at all acceptable
Number of Participants with new or worsening lab abnormalities, Adverse Events (AEs), Serious AEs (SAEs) and AEs Leading to Study Drug Discontinuation in the Double-blind Phase | Up to 48 Weeks
Trough plasma concentration | Baseline, Week 12, Week 24, Week 36, Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Lair, MD, Study Director — Biohaven Pharmaceuticals, Inc.
Locations (53):
- United States (30):
  - Phoenix Children's, Phoenix, Arizona
  - UCSD & Rady Children's, La Jolla, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, Medical Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - UF Health, Shands Hospital, Gainesville, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Northwestern University - Feinberg School of Medicine - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University -Riley Research, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - Boston Children's Hospital - Harvard, Boston, Massachusetts
  - BSHS Office of Research, Grand Rapids, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke University Medicine, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State College of Medicine, Hershey, Pennsylvania
  - CHOP Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Pediatric Neurosciences/Dell Children's Medical Center, Austin, Texas
  - Neurology Rare Disease Center, Denton, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - MultiCare Institute of Research and Innovation, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - University Hospital Antwerp, Edegem
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Leuven
- Czechia (2):
  - University Hospital Brno - Dept. of Pediatric Neurology, Brno
  - Motol University Hospital, Prague
- Germany (3):
  - University Hospital Essen (Public-Law Institution) - Dept. of Pediatrics I, Essen
  - University Hospital Freiburg, Center For Children and Adolescent Medicine, Dept. of Neuropediatrics and Muscle Disorders, Freiburg im Breisgau
  - Dr. Von Haunersches Children'S Hospital - Lmu Munich, Munich
- Italy (4):
  - Irccs Institute of Neurological Sciences of Bologna - Bellaria Hospital, Bologna
  - Nemo-Brescia Clinical Center For Neuromuscular Diseases, Gussago
  - IRCCS NEUROLOGICAL INSTITUTE C. MONDINO CHILD and NEUROPSYCHIATRIC UNIT, Pavia
  - Bambino Gesù Children'S Research Hospital Irccs - San Paolo Office Dept. of Neuroscience, Roma
- University Medical Center Utrecht, Utrecht, Netherlands
- Poland (4):
  - University Clinical Centre in Gdansk - Dept. of Developmental Neurology, Gdansk
  - Heliodor Swiecicki Clinical Hospital At Medical University - Child and Adolescents Neurology Clinic, Poznan
  - The Children'S Memorial Health Institute - Dept. of Neurology and Epileptology, Warsaw
  - T. Marciniak Lower Silesian Specialist Hospital, Pediatric Neurology Dept., Wroclaw
- Spain (4):
  - Donostia University Hospital, Donostia / San Sebastian
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Maternal-Child'S Hospital of Málaga, Regional University Hospital - Pediatric Neurology Unit, Málaga
  - La Fe University and Polytechnic Hospital, Valencia
- United Kingdom (2):
  - Royal Hospital For Children, Glasgow, Scotland
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No